CLINICAL TRIAL: NCT02782455
Title: Calcium Dobesilate vs Flavonoids for the Treatment of Early Hemorrhoidal Disease a Randomised Triple Blind Controlled Trial
Brief Title: Calcium Dobesilate vs Flavonoids for the Treatment of Early Hemorrhoidal Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Postgraduate trainee, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DD
Record Dates: First submitted 2016-03-10; First posted 2016-05-25 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Flavonoids; Diosmin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDobi (Experimental): Calcium dobesylate is given in this group
  Interventions: Drug: CDobi
- Flavono (Active Comparator): Flavonoids are given in this group
  Interventions: Drug: Flavonoids

INTERVENTIONS:
Drug: Flavonoids — Daflon is administered
  Other Names: Daflon
  Arms: Flavono
Drug: CDobi — Calcium dobesylate is administered
  Other Names: dobesilate
  Arms: CDobi

SUMMARY:
Haemorrhoids are vascular cushions in the anal canal that help in the control of stool. When inflamed they become pathological and may present with protrusion and bleeding. A randomized, triple blind , controlled study will be conducted to compare the efficacy of calcium dobesilate against flavanoids in the management of early haemorrhoidal disease.

ELIGIBILITY:
Inclusion Criteria:

* Grade I and Grade II hemorrhoids

Exclusion Criteria:

* CLD
* colorectal/ anorectal Malignancy
* self medication
* local Quack Hakeem medication
* pregnancy

Ages: 13 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Frequency of occurrence of rectal bleeding after usage of drug | 1 weeks
  After the patients will be given the two drugs they will be followed for the frequency of occurrence of rectal bleeding till two weeks

SECONDARY OUTCOMES:
regression of hemorrhoids | 1 weeks
  Patients will under gone per rectal examination and proctoscopy to look for grades of hemorrhoids whether its has decreased or increased.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Waris Farooka, MBBS, FCPS, FRCS, FACS, Study Director — Services Institute of Medical Sciences
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided